CLINICAL TRIAL: NCT03885258
Title: Melatonin Replacement Therapy Effects on Cardiac Autonomic Activity in Pinealectomized Patients
Brief Title: Melatonin Replacement Therapy in Pinealectomized Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ovidiu Constantin Baltatu, Co-PI to PI - José Cipolla-Neto, Anhembi Morumbi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30460114.5.0000.0068
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Pineal Tumor
Keywords: melatonin; pinealectomy; Cardiac Autonomic System; heart rate variability
MeSH Terms: conditions — Pinealoma

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm, single-center, proof-of-concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melatonin Replacement Therapy (Experimental): Melatonin (Aché Pharmaceutics, Brazil) 3 mg, administered in the evening, 30 minutes before the usual bedtime, every day for 3 months. After discontinuation of melatonin therapy, patients are followed up for 6 months to assess safety parameters and cardiac autonomic activity.
  Interventions: Drug: Melatonin Replacement Therapy

INTERVENTIONS:
Drug: Melatonin Replacement Therapy — Melatonin (Aché Pharmaceutics, Brazil), 3 mg, administered in the evening, 30 minutes before the usual bedtime, every day for 3 months. After discontinuation of melatonin therapy, patients are followed up for 6 months to assess safety parameters and cardiac autonomic activity.

SUMMARY:
This is an open-label, single-arm, single-center, proof-of-concept study to assess the effects of melatonin on cardiac autonomic activity in melatonin non-proficient pinealectomized patients.

DETAILED DESCRIPTION:
This is an open-label, single-arm, single-center, proof-of-concept study to assess the effects of melatonin on cardiac autonomic activity in melatonin non-proficient pinealectomized patients. The study consists of a screening period, followed by a 3-month melatonin treatment period, and a 6-month washout follow-up period. Adverse events were monitored with respect to seriousness, intensity, relationship to treatment, action taken and outcome of the event.

ELIGIBILITY:
Inclusion Criteria:

* patients with pinealectomy and all of the following criteria were considered for admission to the clinical trial:
* children, adolescents and young adults 0 months to 25 years of age;
* signed written informed consent (patient or his/her parents/legal guardian);
* willing and able to complete the clinical trial procedures, as described in the protocol
* no recurring tumor after pinealectomy and subsequent chemotherapy
* absence of circulating melatonin evaluated by salivary melatonin Elisa assay

Exclusion Criteria:

* patients with cardiac arrhythmias
* potentially non-compliant subjects judged by the investigator to be unsuitable for the study

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
cardiac autonomic function - heart rate variability | 9 months
  The cardiac autonomic function was determined through heart rate variability (HRV) measures after polysomnography ECG recordings.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cipolla-Neto J, Amaral FGD. Melatonin as a Hormone: New Physiological and Clinical Insights. Endocr Rev. 2018 Dec 1;39(6):990-1028. doi: 10.1210/er.2018-00084. PMID 30215696
- [Background] Baltatu OC, Amaral FG, Campos LA, Cipolla-Neto J. Melatonin, mitochondria and hypertension. Cell Mol Life Sci. 2017 Nov;74(21):3955-3964. doi: 10.1007/s00018-017-2613-y. Epub 2017 Aug 8. PMID 28791422
- [Background] Campos LA, Cipolla-Neto J, Michelini LC. Melatonin modulates baroreflex control via area postrema. Brain Behav. 2013 Mar;3(2):171-7. doi: 10.1002/brb3.123. Epub 2013 Feb 17. PMID 23531786
- [Background] Pereira VL Jr, Dobre M, Dos Santos SG, Fuzatti JS, Oliveira CR, Campos LA, Brateanu A, Baltatu OC. Association between Carotid Intima Media Thickness and Heart Rate Variability in Adults at Increased Cardiovascular Risk. Front Physiol. 2017 Apr 26;8:248. doi: 10.3389/fphys.2017.00248. eCollection 2017. PMID 28491040
- [Background] Campos LA, Pereira VL Jr, Muralikrishna A, Albarwani S, Bras S, Gouveia S. Mathematical biomarkers for the autonomic regulation of cardiovascular system. Front Physiol. 2013 Oct 7;4:279. doi: 10.3389/fphys.2013.00279. PMID 24109456
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Derived] Campos LA, Bueno C, Barcelos IP, Halpern B, Brito LC, Amaral FG, Baltatu OC, Cipolla-Neto J. Melatonin Therapy Improves Cardiac Autonomic Modulation in Pinealectomized Patients. Front Endocrinol (Lausanne). 2020 Apr 30;11:239. doi: 10.3389/fendo.2020.00239. eCollection 2020. PMID 32431667